CLINICAL TRIAL: NCT01013389
Title: A Prospective, Randomised Study Comparing the Use of Actifuse (Trademark)ABX Synthetic Bone Substitute With INFUSE (Registrered Trademark) in Patients Requiring Posterolateral Instrumented Lumbar Fusion With Interbody Fusion
Brief Title: Actifuse ABX Versus INFUSE in Posterolateral Instrumented Lumbar Fusion (PLIF) With Interbody Fusion
Acronym: APPRAISET1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Collaborators: Apatech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIP0702PLF; ACTRN12609000527268; EudraCT Number: 2009-012672-27
Record Dates: First submitted 2009-11-10; First posted 2009-11-13 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Degenerative Disc Disease
Keywords: actifuse; INFUSE; InductOs; DDD; degenerative disk disease; PLIF; PITF; PLF; poterolateral lumber fusion; Bone substitute; bone graft; synthetic bone substitute
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Actifuse ABX (Experimental): Actifuse ABX bone substitute
  Interventions: Procedure: Actifuse ABX
- INFUSE, plus master granules (MGG) (Active Comparator): synthetic bone substitute used in posterolateral instrumented lumber fusion with interbody fusion
  Interventions: Procedure: INFUSE, plus master granules (MGG)

INTERVENTIONS:
Procedure: Actifuse ABX — bone substitute used for posterolateral instrumented lumbar fusion with interbody fusion
  Arms: Actifuse ABX
Procedure: INFUSE, plus master granules (MGG) — bone substitute in posterolateral instrumented lumbar fusion with interbody fusion
  Arms: INFUSE, plus master granules (MGG)

SUMMARY:
The primary objective of this clinical trial is to evaluate the success rates of Actifuse ABX and INFUSE in achieving bone fusion.

The secondary objective of this clinical trial is to assess clinical outcome measurements.

ELIGIBILITY:
Inclusion Criteria:

* Has degenerative disc disease of the lumbar spine as indicated by back pain of discogenic/degenerative origin, with or without leg pain, and has one or more of the following conditions as documented by plain X-rays, CT scan or MRI scan:

  * Modic changes.
  * High intensity changes in the annulus.
  * Loss of disc height.
  * Decreased hydration of the disc.
  * Canal stenosis with or without spondylotic slip.
  * Gross facet joint changes requiring fusion for treatment.
  * Have documented annular pathology by other means. (e.g., with discography).
* Has a preoperative Oswestry Back Disability Score of 30 or more.
* Aged 18 to 75 years and skeletally mature at time of surgery.
* Has not responded to non-operative treatment (e.g., bed rest, physical therapy, medications and/or spinal injections) for a period of six months.
* If of childbearing potential, patient is non-pregnant, non-nursing and agrees not to become pregnant for one year following surgery.
* Is willing to and able to comply with the study plan and able to understand and sign the Patient Informed Consent Form.

Exclusion Criteria:

* Has had previous failed attempts at fusion surgery at the involved level(s).
* Has a diagnosis of spinal infection tumour or trauma.
* Requires surgery at more than two (2) levels.
* Has osteoporosis (excluding osteopenia) as evidenced on plain X-rays, CT scans (or DEXA scan in cases of doubt).
* Is pregnant.
* Is an alcohol and/or drug abuser as defined by currently undergoing treatment for alcohol and/or drug abuse.
* Has received drugs that may interfere with bone metabolism within two weeks prior to the planned surgery date (e.g., steroids or methotrexate) excluding routine perioperative, non-steroidal anti-inflammatory drugs.
* Has a history of autoimmune disease.
* Has a history of exposure to injectable collagen implants.
* Has a history of hypersensitivity to protein pharmaceuticals (monoclonal antibodies or gamma globulins) or collagen.
* Has received treatment with an investigational therapy (device and/or pharmaceutical) within 30 days prior to surgery or such treatment is planned during the 24 months following surgery.
* Has received any previous exposure to any/all BMPs of either human or animal extraction.
* Has a history of allergy to bovine products or a history of general anaphylaxis.
* Has a history of any endocrine or metabolic disorder known to affect osteogenesis (e.g., Paget's disease, renal oseodystrophy, Ehlos-Danlos syndrome or osteogenesis imperfecta).
* Has any disease that would preclude accurate clinical evaluation (e.g., neuromuscular disease, etc.).
* Has a primary diagnosis of a spinal disorder other than degenerative disc disease or other conditions as set out in "inclusions" above at the involved level(s).
* Has a condition that requires postoperative medications that interfere with fusion, such as steroids or prolonged use of non-steroidal anti-inflammatory drugs, excluding routine perioperative non-steroidal anti-inflammatory drugs. This does not include low dose aspirin for prophylactic anticoagulation.
* Has overt or active bacterial infection, local or systemic, and/or a potential for bacteremia.
* Has presence of active malignancy or prior history of malignancy (except for basal cell carcinoma of the skin).
* Has a documented metal allergy or intolerance to titanium alloy or cobalt-chrome-molybdenum alloy.
* Is, in the opinion of the Principal Investigator or Co-Investigators, intellectually unable to co-operate with the study.
* Has chronic or acute renal and/or hepatic failure or prior history of renal or hepatic disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Fusion, defined as evidence of bridging trabecular bone present at 1 year as assessed by CT scan as well as a determination of no motion as assessed by plain radiographs. | 1 year

SECONDARY OUTCOMES:
Improvement clinical outcomes measurements compared to pre-opscores: pain/Disability as measured by Oswestry Lower Back Pain Questionnaire, quality of Life as measured by Short Form Health Survey (SF36), and neurological status | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Huub Kreuwel, Ph.D, Study Director — Director, Medical Affairs
Locations (2):
- Moloney & Associates, Wollongong, Australia
- Isala Klinik, Zwolle, Netherlands